CLINICAL TRIAL: NCT04039763
Title: Assessment of the Impact of Real-time Continuous Glucose Monitoring on Glycaemic Control in High-risk Adolescents and Young Adults With Insulin-treated Diabetes
Brief Title: RT-CGM in Young Adults at Risk of DKA
Acronym: YODA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19SM5161
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Disease; Autoimmune Diseases; Endocrine System Diseases
Keywords: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Autoimmune Diseases; Endocrine System Diseases | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Randomised controlled crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Real Time Continuous Glucose Monitoring (Experimental): Participants wear Real time continous glucose monitoring (Dexcom G6), with alarms for when their glucose is too low or too high. They will be able to view their data on the Dexcom app on their smartphones or a Dexcom receiver and share this with a nominated caregiver. Participants can chose to share data between study visits via "Dexcom clarity" with the research/clinical team, who will support them making changes to their insulin regime in light of the data.
  Interventions: Device: Dexcom G6
- Standard care (Placebo Comparator): Standard care - finger prick self monitoring of blood glucose.
  Interventions: Device: Self monitoring of blood glucose

INTERVENTIONS:
Device: Dexcom G6 — Realtime Continous Glucose Monitoring
  Arms: Real Time Continuous Glucose Monitoring
Device: Self monitoring of blood glucose — Finger prick self monitoring of blood glucose
  Arms: Standard care

SUMMARY:
Pilot study to evaluate the effect of real time continuous glucose monitoring (RT-CGM) on young-adults with insulin-treated diabetes, who are defined as high risk due to suboptimal HbA1c (blood glucose control) or a history of hospital admissions for high blood glucoses.

Hypothesis: RT-CGM provided to young adults with suboptimal blood glucose control, has a beneficial impact on HbA1c and hospital admissions for high blood glucoses. We will use data from this pilot work to inform a larger powered study to address this knowledge gap.

DETAILED DESCRIPTION:
Real time continous glucose monitoring (RT-CGM) is a technology that measures people's sugar level all the time, using a sensor that is placed on the skin. The sensor can be worn for 10 days and the small transmitter clicks into the sensor and sends the glucose readings wirelessly to a smartphone or a small handset, which displays the glucose level on the screen. It also has alarms to tell people when their sugar level is too high or too low. This study uses the Dexcom G6 RT-CGM system.

RT-CGM devices have become smaller and can connect easily with mobile phones. We want to find out whether young people, in particular, find the technology useful and whether it improves how they self-managed their diabetes over a 6-month period.

This is a randomised controlled cross over trial; participants are randomly assigned to the control group (standard care which is self-monitoring of blood glucose via fingerprick) or the intervention group (RT-CGM) for the first 6 months and then cross over for the 2nd 6 months. Participants will be able to share their CGM data if they wish via Dexcom Clarity with the research/clinical team, who will support them in making treatment decisions in light of the data.

All participants will be asked to take part in a semi-structured interview with a Diabetes Specialist Clinical Psychologist at baseline, including to address some of the barriers to self-management and a further interview at the end of the 6 months during which they use RT- CGM, to explore their experiences using it. All participants will be asked to complete validated psychology questionnaires at baseline, 6 months and 12 months. A blood test for HbA1C will be done at baseline, 6 months and 12 months. After 12 months, all participants will be invited to attend a focus group to provide feedback & share their experiences of using RT-CGM and raise themes brought up in psychology interviews to the whole group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults aged 18-25 years
* Insulin-treated diabetes >12 months (on multiple daily injections or insulin pump therapy)
* HbA1c > 75 mmol/mol (9%) or 1 or more DKA admissions in the last 12 months or 1 or more admissions with uncontrolled blood glucose levels in the last 12 months.
* Naïve to RT-CGM - except for short periods for use for diagnosis or monitoring purposes.
* Use of prior flash glucose monitoring is permittable

Exclusion Criteria:

* Chronic kidney disease eGFR <30ml/min
* Pregnant or planning pregnancy
* Breastfeeding
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Unable to participate due to other factors, as assessed by the Chief Investigator

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haeomglobin (HbA1c) | Over 6 months for intervention period and over 6 months for control period (total 12 months)
  Change over intervention period or standard care (control) period, with each participant acting as their own control

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Misra, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No